CLINICAL TRIAL: NCT02346188
Title: Effects of Iron and Zinc Supplementation on Neuropsychological and Educational Achievement in Lead-exposed School Children
Brief Title: Effects of Iron and/or Zinc Supplementation in Mexican School Children Exposed to Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other); National Polytechnic Institute, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H.22.00.07.06B
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Lead Poisoning
Keywords: blood lead, iron, zinc, child, cognition, behavior, Mexico
MeSH Terms: conditions — Lead Poisoning; Behavior | interventions — ferrous fumarate; Zinc Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ferrous fumarate (Experimental): Tablet formulated as ferrous fumarate, 30 mg. Given once daily for 6 months.
  Interventions: Dietary Supplement: Ferrous fumarate
- Zinc oxide (Experimental): Tablet formulated as zinc oxide, 30 mg. Given once daily by mouth for 6 months.
  Interventions: Dietary Supplement: Zinc oxide
- Ferrous fumarate and zinc oxide (Experimental): Tablet, formulated as ferrous fumarate 30 mg plus zinc oxide 30 mg. Given once daily by mouth for 6 months.
  Interventions: Dietary Supplement: Ferrous fumarate; Dietary Supplement: Zinc oxide
- Placebo (Placebo Comparator): Sugar tablet formulated to look like the experimental arms of the study. Given daily by mouth for 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ferrous fumarate — Tablet formulated from 30 mg ferrous fumarate.
  Arms: Ferrous fumarate; Ferrous fumarate and zinc oxide
Dietary Supplement: Zinc oxide — Tablet formulated from 30 mg zinc oxide
  Arms: Ferrous fumarate and zinc oxide; Zinc oxide
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Lead is negatively linked to nutritional status, behavior and cognition in children. Despite extensive knowledge of its toxicity and efforts to reduce exposure, lead continues to be a problem in developed and developing countries. When lead exposure is unavoidable due to its pervasive nature, effective means of protecting or disrupting that exposure need to be developed. Nutritional interventions are one such option. We conducted a 2x2 factorial, placebo-controlled trial of 6-month iron and zinc supplementation among lead-exposed children in Torreón, Mexico (altitude 1060 m). Nine schools were selected based on proximity to a lead smelter and first-graders were individually randomized to daily treatment with 30 mg iron, 30 mg zinc, both, or placebo. In addition to biochemical indicators, cognitive functions and behavior were evaluated at baseline, after the 6-month supplementation period, and again after another 6 months (without supplementation).

At baseline, 602 children ages 6.2-8.5 years were enrolled.

DETAILED DESCRIPTION:
We conducted a 2x2 factorial, placebo-controlled trial of 6-month iron and zinc supplementation among lead-exposed children in Torreón, Mexico (altitude 1060 m) to test the hypothesis that supplementation with iron, zinc or both will reduce blood lead concentrations of the children and improve their cognition and behavior. Nine schools were selected based on proximity to a lead smelter and first-graders were individually randomized to daily treatment with 30 mg iron, 30 mg zinc, both, or placebo. In addition to biochemical indicators (blood lead, serum ferritin, CRP, serum zinc, urinary arsenic concentrations), cognitive functions and behavior were measured. Assessments were conducted at three time points: at baseline, after the 6 month treatment, and again after another 6 months without treatment. At baseline, 602 children ages 6.2-8.5 years were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1st grade child

Exclusion Criteria:

* Blood lead concentration =>45 ug/dL
* Hemoglobin concentration < 9 g/dL

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 602 (Actual)
Dates: Start 2000-01; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Blood lead concentration | 6-12 months

SECONDARY OUTCOMES:
Anthropometric composite | 6-12 months
  Height, weight
Serum ferritin concentration | 6-12 months
Serum zinc concentration | 6-12 months
Hemoglobin concentration | 6-12 months
Conners Behavior Rating Scales for parents and teachers | 6-12 months
Peabody Picture Vocabulary Test, Math achievement test, tests of attention and memory | 6-12 months

OTHER OUTCOMES:
Arsenic exposure | 6-12 months
  total urinary arsenic, inorganic arsenic, monomethylarsonic acid, dimethylarsinic acid

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Stoltzfus, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Result] Kordas K, Lopez P, Rosado JL, Garcia Vargas G, Alatorre Rico J, Ronquillo D, Cebrian ME, Stoltzfus RJ. Blood lead, anemia, and short stature are independently associated with cognitive performance in Mexican school children. J Nutr. 2004 Feb;134(2):363-71. doi: 10.1093/jn/134.2.363. PMID 14747673
- [Result] Kordas K, Canfield RL, Lopez P, Rosado JL, Vargas GG, Cebrian ME, Rico JA, Ronquillo D, Stoltzfus RJ. Deficits in cognitive function and achievement in Mexican first-graders with low blood lead concentrations. Environ Res. 2006 Mar;100(3):371-86. doi: 10.1016/j.envres.2005.07.007. Epub 2005 Sep 19. PMID 16169549
- [Result] Kordas K, Stoltzfus RJ, Lopez P, Rico JA, Rosado JL. Iron and zinc supplementation does not improve parent or teacher ratings of behavior in first grade Mexican children exposed to lead. J Pediatr. 2005 Nov;147(5):632-9. doi: 10.1016/j.jpeds.2005.06.037. PMID 16291354
- [Result] Rico JA, Kordas K, Lopez P, Rosado JL, Vargas GG, Ronquillo D, Stoltzfus RJ. Efficacy of iron and/or zinc supplementation on cognitive performance of lead-exposed Mexican schoolchildren: a randomized, placebo-controlled trial. Pediatrics. 2006 Mar;117(3):e518-27. doi: 10.1542/peds.2005-1172. PMID 16510631
- [Result] Rosado JL, Lopez P, Kordas K, Garcia-Vargas G, Ronquillo D, Alatorre J, Stoltzfus RJ. Iron and/or zinc supplementation did not reduce blood lead concentrations in children in a randomized, placebo-controlled trial. J Nutr. 2006 Sep;136(9):2378-83. doi: 10.1093/jn/136.9.2378. PMID 16920858
- [Result] Rosado JL, Ronquillo D, Kordas K, Rojas O, Alatorre J, Lopez P, Garcia-Vargas G, Del Carmen Caamano M, Cebrian ME, Stoltzfus RJ. Arsenic exposure and cognitive performance in Mexican schoolchildren. Environ Health Perspect. 2007 Sep;115(9):1371-5. doi: 10.1289/ehp.9961. PMID 17805430
- [Result] Kordas K, Casavantes KM, Mendoza C, Lopez P, Ronquillo D, Rosado JL, Vargas GG, Stoltzfus RJ. The association between lead and micronutrient status, and children's sleep, classroom behavior, and activity. Arch Environ Occup Health. 2007 Summer;62(2):105-12. doi: 10.3200/AEOH.62.2.105-112. PMID 18316268
- [Result] Roy A, Kordas K, Lopez P, Rosado JL, Cebrian ME, Vargas GG, Ronquillo D, Stoltzfus RJ. Association between arsenic exposure and behavior among first-graders from Torreon, Mexico. Environ Res. 2011 Jul;111(5):670-6. doi: 10.1016/j.envres.2011.03.003. Epub 2011 Mar 25. PMID 21439564
- [Result] Moodie S, Ialongo N, Lopez P, Rosado J, Garcia-Vargas G, Ronquillo D, Kordas K. The conjoint influence of home enriched environment and lead exposure on children's cognition and behaviour in a Mexican lead smelter community. Neurotoxicology. 2013 Jan;34:33-41. doi: 10.1016/j.neuro.2012.10.004. Epub 2012 Oct 27. PMID 23110976
- [Derived] Kordas K, Roy A, Lopez P, Garcia-Vargas G, Cebrian ME, Vera-Aguilar E, Rosado JL. Iron and Zinc Supplementation Does Not Impact Urinary Arsenic Excretion in Mexican School Children. J Pediatr. 2017 Jun;185:205-210.e1. doi: 10.1016/j.jpeds.2017.02.040. Epub 2017 Mar 23. PMID 28343659